CLINICAL TRIAL: NCT05817227
Title: Selenoproteins as Prognostic Markers and Therapeutic Targets in Breast Cancer.
Acronym: Selebrec
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: SELEBREC; 57/21oss (Other: IRCCS I.N.T. "G. Pascale")
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is multicentric, spontaneous, observational, retrospective and prospective study.

DETAILED DESCRIPTION:
In the retrospective part of the study, Tissue Microarrays (TMA) will be prepared from surgical samples of breast tissue from a series of patients with TNBC type breast cancer.

In the prospective part of the study will be evaluated the expression of some selenoproteins by ELISA in plasma samples obtained from up to 100 healthy subjects and about 300 (~100 per year) patients with basally metastatic TNBC breast cancer (150) and metastatic (150) before any treatment.

ELIGIBILITY:
Inclusion Criteria:

* TNBC breast cancer patients, before any drug treatment
* healthy women aged 25-60

Exclusion Criteria:

* donors suffering from diabetes, hypertension, active infectious states, HIV infection, Hepatitis B or C, chronic inflammatory diseases, current or previous neoplasms, heart disease or drug treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients included in the study are all women and have an age below 40 in 26/235 (11.1%) cases, between 40 and 60 in 108/235 (46.0%) cases and over 60 for 101/235 (43.0%) cases.
  Tumours have the following clinical and pathological characteristics: 204/235 (86.8%) are carcinomiducts and 31/235 (13.2%) are non ductal carcinomas; 202/235 (86%) grade 3, 31/235 (13.1%) grade 2 and 2/235 (0.9%) grade 1; tumour dimensions are less than 2 cm (T1) in 103/225 cases (45.8%), between 2 and 5 cm in 103/225 (45.8%) and greater than 5 cm in 19/225 (8.4%). Expression of Ki67 diproliferation factor was high (>20%) in 186/227 (81.9%) patients and low (<20%) in 41/227 (18.1%). At the date of surgery 97/232 (41.8%) patients had lymphonode metastases, while 44/111 (39.6%) had distant metastases.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2027-11-19 (Estimated); Study Completion 2027-11-19 (Estimated)

PRIMARY OUTCOMES:
Use of immunohistochemistry investigation (IHC) | 3 years
  In the retrospective part of the study, Tissue Microarrays (TMA) will be prepared from surgical samples of breast tissue from a series of patients with TNBC type breast cancer. The expression of some of the twenty-five selenoproteins will be evaluated by immunohistochemical investigation (IHC) on the TMA (Tumor Microarrays).
Prospective evaluation of expression of some selenoproteins by kit ELISA in plasma samples | 3 years
  In the prospective part of the study will be evaluated the expression of some selenoproteins by ELISA in plasma samples obtained from up to 100 healthy subjects and about 300 (~100 per year) patients with basally metastatic TNBC breast cancer (150) and metastatic (150) before any treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Budillon, M.D., Principal Investigator — IRCCS I.N.T. "G. Pascale"; Susan Costantini, PhD, Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (2):
- Italy (2):
  - Istituto Nazionale Tumori - Fondazione "G.Pascale", IRCCS, Napoli, Napoli
  - Istituto Nazionale Tumori Regina Elena, Roma, Roma

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- [Background] DeSantis CE, Ma J, Gaudet MM, Newman LA, Miller KD, Goding Sauer A, Jemal A, Siegel RL. Breast cancer statistics, 2019. CA Cancer J Clin. 2019 Nov;69(6):438-451. doi: 10.3322/caac.21583. Epub 2019 Oct 2. PMID 31577379
- [Background] Garrido-Castro AC, Lin NU, Polyak K. Insights into Molecular Classifications of Triple-Negative Breast Cancer: Improving Patient Selection for Treatment. Cancer Discov. 2019 Feb;9(2):176-198. doi: 10.1158/2159-8290.CD-18-1177. Epub 2019 Jan 24. PMID 30679171
- [Background] Lu J, Holmgren A. Selenoproteins. J Biol Chem. 2009 Jan 9;284(2):723-7. doi: 10.1074/jbc.R800045200. Epub 2008 Aug 29. PMID 18757362
- [Background] Short SP, Williams CS. Selenoproteins in Tumorigenesis and Cancer Progression. Adv Cancer Res. 2017;136:49-83. doi: 10.1016/bs.acr.2017.08.002. PMID 29054422
- [Background] Marciel MP, Hoffmann PR. Selenoproteins and Metastasis. Adv Cancer Res. 2017;136:85-108. doi: 10.1016/bs.acr.2017.07.008. Epub 2017 Sep 1. PMID 29054423
- [Background] Avery JC, Hoffmann PR. Selenium, Selenoproteins, and Immunity. Nutrients. 2018 Sep 1;10(9):1203. doi: 10.3390/nu10091203. PMID 30200430
- [Background] Varlamova EG. Participation of selenoproteins localized in the ER in the processes occurring in this organelle and in the regulation of carcinogenesis-associated processes. J Trace Elem Med Biol. 2018 Jul;48:172-180. doi: 10.1016/j.jtemb.2018.04.005. Epub 2018 Apr 3. PMID 29773177
- [Background] Guariniello S, Di Bernardo G, Colonna G, Cammarota M, Castello G, Costantini S. Evaluation of the selenotranscriptome expression in two hepatocellular carcinoma cell lines. Anal Cell Pathol (Amst). 2015;2015:419561. doi: 10.1155/2015/419561. Epub 2015 Jun 23. PMID 26199857
- [Background] Capone F, Polo A, Sorice A, Budillon A, Costantini S. Integrated Analysis to Study the Relationship between Tumor-Associated Selenoproteins: Focus on Prostate Cancer. Int J Mol Sci. 2020 Sep 13;21(18):6694. doi: 10.3390/ijms21186694. PMID 32933107
- [Background] Lopez-Saez JB, Senra-Varela A, Pousa-Estevez L. Selenium in breast cancer. Oncology. 2003;64(3):227-31. doi: 10.1159/000069312. PMID 12697962
- [Background] Debski MG, Pachucki J, Ambroziak M, Olszewski W, Bar-Andziak E. Human breast cancer tissue expresses high level of type 1 5'-deiodinase. Thyroid. 2007 Jan;17(1):3-10. doi: 10.1089/thy.2006.0012. PMID 17274741
- [Background] Cha MK, Suh KH, Kim IH. Overexpression of peroxiredoxin I and thioredoxin1 in human breast carcinoma. J Exp Clin Cancer Res. 2009 Jun 30;28(1):93. doi: 10.1186/1756-9966-28-93. PMID 19566940
- [Background] Pellatt AJ, Wolff RK, John EM, Torres-Mejia G, Hines LM, Baumgartner KB, Giuliano AR, Lundgreen A, Slattery ML. SEPP1 influences breast cancer risk among women with greater native american ancestry: the breast cancer health disparities study. PLoS One. 2013 Nov 20;8(11):e80554. doi: 10.1371/journal.pone.0080554. eCollection 2013. PMID 24278290
- [Background] Ravn-Haren G, Olsen A, Tjonneland A, Dragsted LO, Nexo BA, Wallin H, Overvad K, Raaschou-Nielsen O, Vogel U. Associations between GPX1 Pro198Leu polymorphism, erythrocyte GPX activity, alcohol consumption and breast cancer risk in a prospective cohort study. Carcinogenesis. 2006 Apr;27(4):820-5. doi: 10.1093/carcin/bgi267. Epub 2005 Nov 14. PMID 16287877
- [Background] Hu YJ, Diamond AM. Role of glutathione peroxidase 1 in breast cancer: loss of heterozygosity and allelic differences in the response to selenium. Cancer Res. 2003 Jun 15;63(12):3347-51. PMID 12810669
- [Background] Knight JA, Onay UV, Wells S, Li H, Shi EJ, Andrulis IL, Ozcelik H. Genetic variants of GPX1 and SOD2 and breast cancer risk at the Ontario site of the Breast Cancer Family Registry. Cancer Epidemiol Biomarkers Prev. 2004 Jan;13(1):146-9. doi: 10.1158/1055-9965.epi-03-0164. PMID 14744747
- [Background] Rusolo F, Capone F, Pasquale R, Angiolillo A, Colonna G, Castello G, Costantini M, Costantini S. Comparison of the seleno-transcriptome expression between human non-cancerous mammary epithelial cells and two human breast cancer cell lines. Oncol Lett. 2017 Apr;13(4):2411-2417. doi: 10.3892/ol.2017.5715. Epub 2017 Feb 13. PMID 28454412
- [Background] Nunziata C, Polo A, Sorice A, Capone F, Accardo M, Guerriero E, Marino FZ, Orditura M, Budillon A, Costantini S. Structural analysis of human SEPHS2 protein, a selenocysteine machinery component, over-expressed in triple negative breast cancer. Sci Rep. 2019 Nov 6;9(1):16131. doi: 10.1038/s41598-019-52718-0. PMID 31695102
- [Background] Costantini S, Capone F, Polo A, Bagnara P, Budillon A. Valosin-Containing Protein (VCP)/p97: A Prognostic Biomarker and Therapeutic Target in Cancer. Int J Mol Sci. 2021 Sep 21;22(18):10177. doi: 10.3390/ijms221810177. PMID 34576340
- [Background] Epplein M, Burk RF, Cai Q, Hargreaves MK, Blot WJ. A prospective study of plasma Selenoprotein P and lung cancer risk among low-income adults. Cancer Epidemiol Biomarkers Prev. 2014 Jul;23(7):1238-44. doi: 10.1158/1055-9965.EPI-13-1308. Epub 2014 Apr 24. PMID 24762559
- [Background] Yu SS, Du JL. Selenoprotein S: a therapeutic target for diabetes and macroangiopathy? Cardiovasc Diabetol. 2017 Aug 10;16(1):101. doi: 10.1186/s12933-017-0585-8. PMID 28797256